CLINICAL TRIAL: NCT02833623
Title: Efficacy of Short-message-based Re-education (SMRE) on Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016SDU-QILU-07
Record Dates: First submitted 2016-07-07; First posted 2016-07-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Helicobacter Pylori Eradication Rate
Keywords: Helicobacter Pylori eradication rate; Efficacy of Short-message-based Re-education (SMRE)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short-message-based Re-education group (Experimental): Patients receive oral and written education before H. pylori eradication therapy at first, then they receive short message re-education twice per day during therapy.
  Both the content of the oral and written education and the short message re-education are same.
  Interventions: Behavioral: Short-message-based Re-education
- conventional education group (Active Comparator): Patients only receive oral and written education before H. pylori eradication therapy.
  Interventions: Behavioral: conventional education

INTERVENTIONS:
Behavioral: Short-message-based Re-education
  Arms: Short-message-based Re-education group
Behavioral: conventional education
  Arms: conventional education group

SUMMARY:
Helicobacter pylori (H. pylori) is a pathogen that infects more than 50% of the human population, resulting in high healthcare costs worldwide. However, H. pylori eradication rate is low nowadays and patients's compliance is one of the most important effective factors.

ELIGIBILITY:
Inclusion Criteria:

* outpatients aged 18-70 years
* confirmed diagnosis of H. pylori infection by at least one of the following methods: 13C-urea breath test, histology, rapid urease test or bacterial culture
* an intention of H. pylori eradication treatment and have written inform consent
* ability to read short messages on the mobile phone

Exclusion Criteria:

* advanced chronic disease that would not allow the patient to complete the treatment or follow-up or attend visits
* allergy to any of the drugs used in this study
* previous Helicobacter Pylori eradication treatment
* pregnancy or breastfeeding (female participants with childbearing potential were required to use medically accepted contraception for the duration of the study)
* taking antibiotics or PPIs or bismuth salts within four weeks
* previous gastrointestinal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The difference of H. pylori eradication rate between two groups | 8 months

SECONDARY OUTCOMES:
Rate of non-compliance with instructions between 2 groups | 8 months

OTHER OUTCOMES:
The different rate of adverse events between 2 groups | 8 months
The different rate of symptom remissions after Hp eradication therapy between 2 groups | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China